CLINICAL TRIAL: NCT00639522
Title: A Phase I Clinical Trial to Investigate the Maximum Tolerated Dose and Pharmacokinetics of Liposomal Paclitaxel With/Without Capecitabine in Chinese Cancer Patients With Advanced Gastric Carcinoma.
Brief Title: Dose Escalation Study of Liposomal Paclitaxel With/Without Capecitabine in Patients With Advanced Gastric Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Prof. Jinwan Wang, Cancer Institute and Hospital,Chinese Academy of Medical Science
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS-GC-01-2008
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Gastric Carcinoma
Keywords: Liposomal paclitaxel; Maximum tolerated dose; Pharmacokinetics; Gastric carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Liposomal paclitaxel and capecitabine

INTERVENTIONS:
Drug: Liposomal paclitaxel and capecitabine — Patients will be given Liposomal paclitaxel intravenously in 3 hours with the dose of 175mg/m2、185mg/m2、195mg/m2、 200mg/m2、205mg/m2 and so on ,at the first day of chemotherapy. Capecitabine will be given on d1 to d14 with the dose of 185mg/m2、200mg/m2 or d8 to d21 with the dose of 175mg/m2、195mg/m2、205mg/m2 .Cycle duration will be 21 days. Each patient will receive 2 cycles of therapy. Only in the first cycle blood samples will be taken on 16 points in 48 hours after the infusion of liposomal paclitaxel.

SUMMARY:
The purpose of this study is to investigate the maximum tolerated dose and pharmacokinetics of liposomal paclitaxel with/without capecitabine in Chinese cancer patients with advanced gastric carcinoma.

DETAILED DESCRIPTION:
The maximum tolerated dose (MTD) and pharmacokinetics of a new formulation of taxane (liposomal paclitaxel) have never been studied in Chinese cancer patients, either alone or with capecitabine .This clinical trial is designed to find out the MTD and pharmacokinetics of liposomal paclitaxel with a beginning dose of 175mg/m2 with/without Capecitabine in Chinese patients with advanced gastric carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified gastric carcinoma of advanced stages which is unsuitable for surgery;
* No prior systemic chemotherapy with taxane at least 6 months before the recruitment;
* At least one measurable tumor according to RECIST standard, with at least one diameter ≥20mm assessed by traditional imaging technique or MRI, or with a diameter twice of the thickness of scan layer (or ≥10-16mm) under spiral CT; Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
* Patients who are expected to live at least 3 months;
* Obtaining informed consent;

Exclusion Criteria:

* Receiving other chemotherapy or radiotherapy during the administration;
* Symptomatic metastatic brain tumor;
* Allergy to any study medication;
* Pregnancy or breast feeding;
* Severe heart diseases;
* Uncontrolled mental diseases;
* Abnormal liver and renal functions, which are measured by AST/ALT and BUN/Cr;
* Neutrophils（ANC）<2000/μL;platelets<100，000/μL;hemoglobin（HB）<9.0 g/dL;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | 6 weeks

SECONDARY OUTCOMES:
Pharmacokinetics | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, Doctor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital,Chinese Academy of Medical Science, Beijing, Beijing Municipality, China